CLINICAL TRIAL: NCT06944548
Title: Evaluation of the Effect of Adapted Physical Activity on the Modification of Lipid Metabolism During Chemotherapy for Metastatic COLorectal Cancer
Acronym: APACOL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A00415-44
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (CRC); Volunteer Subjects
Keywords: No special diet; ECOG 0 or 1; Blood albumin ≥30g/L; Age ≥ 18 years; Patients eligible for chemotherapy treatment
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 - Arms without teacher intervention for adapted physical activity (Active Comparator): For this group:
  * Patient inclusion
  * No adapted physical activity programme set up and no follow-up by an adapted physical activity teacher
  * Collection of daily adapted physical activity via a paper diary for 8 weeks.
  * 3 blood samples for lipidomic analysis
  * Functional physical assessment
  * Completion of various questionnaires: quality of life, previous physical activity and dietary intake
  Interventions: Biological: Lipidomic analyses; Other: Adapted physical activity program
- Group 2 - Arm " intervention by an adapted physical activity teacher - minimum volume of INCa recomm (Active Comparator): For this group:
  * Patient inclusion
  * Implementation of an adapted physical activity programme supervised by a teacher offering 180 minutes of adapted physical activity per week for 8 weeks. Minimum volume recommended by INCa.
  * 3 blood samples for lipidomic analysis
  * Functional physical assessment
  * Completion of various questionnaires: quality of life, previous physical activity and dietary intake
  Interventions: Biological: Lipidomic analyses; Other: Adapted physical activity program
- Group 3 - Arm " intervention by an adapted physical activity teacher - maximum volume of INCa recomm (Active Comparator): For this group:
  * Patient inclusion
  * Implementation of an adapted physical activity programme supervised by a teacher offering 300 minutes of adapted physical activity per week for 8 weeks. Maximum volume per week recommended by INCa.
  * 3 blood samples for lipidomic analysis
  * Functional physical assessment
  * Completion of various questionnaires: quality of life, previous physical activity and dietary intake
  Interventions: Biological: Lipidomic analyses; Other: Adapted physical activity program
- Group 4 - Healthy volunteers (Active Comparator): For this group:
  * Volunteers inclusion
  * 3 blood samples for lipidomic analysis
  * Functional physical assessment
  * Completion of questionnaire : previous physical activity
  Interventions: Biological: Lipidomic analyses; Other: Adapted physical activity program

INTERVENTIONS:
Biological: Lipidomic analyses — 3 blood samples taken from 2 x 6 mL EDTA tubes for patients
  * At baseline
  * Week 5 of the adapted physical activity protocol
  * Follow-up visit for adapted physical activity
    1 blood sample taken from 2 x 6 mL EDTA tubes for volunteers
  * At baseline
Other: Adapted physical activity program — 8-week adapted physical activity program. This program will be adapted to each group

SUMMARY:
APACOL is a pilot, bicentric, randomised, open-label, prospective, category 2 study. The presence of colon cancer modifies blood lipid parameters which are likely to have an impact on the efficacy of anti-cancer treatments. Previous data support the hypothesis that appropriate physical activity could modify the blood lipid parameters involved in chemoresistance in patients with metastatic colorectal cancer.

The aim of the APACOL study is to investigate the impact of modulating the frequency (volume per week) of physical activity recommended by INCa on the variation in lipid parameters involved in chemoresistance in patients with metastatic colon cancer, with a reference level of these lipid parameters in people without cancer provided by the participation of volunteers who are not ill.

The expectations at the end of this study are an improvement in the patient's quality of life / an improvement in the tolerance and efficacy of the chemotherapy treatment / identification of the frequency of APAs needed to vary the lipid metabolism involved in chemoresistance.

DETAILED DESCRIPTION:
This study will be open on 2 sites (CIC CHU Dijon with inclusion of 18 volunteers and CGFL with inclusion of 36 patients).

The participants will be randomized in 4 differents groups :

* Group 1 (for patients only) : No adapted physical activity teacher arm
* Groupe 2 (for patients only) : Arm intervention with an adapted physical activity teacher - minimum volume of INCa recommendations for adapted physical activity
* Groupe 3 (for patients only) : Arm intervention with an adapted physical activity teacher - maximum volume of INCa recommendations for adapted physical activity
* Groupe 4 (for volunteers only) Each participant in the 4 groups will have to complete questionnaires (quality of life, physical activity and dietary intake) and take 3 blood samples for lipidomic analysis.

For patients in groups 1 to 3, participants will be asked to complete a diary to record their daily physical activity and the duration of that activity.

For groups 2 and 3, in addition to the diary, sessions with adapted physical activity teaching will be organised throughout the study.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥ 18 years
* Patient with histologically proven metastatic colorectal cancer
* Patient eligible for treatment with chemotherapy, in combination or not with other anti-cancer treatments according to standard management
* Have a performance status of 0 or 1 according to the WHO ECOG index
* Blood albumin value ≥30g/L
* Patient able to give consent and able to undergo study monitoring, including visits, physical activities, blood sampling
* Patient affiliated to a social security scheme or equivalent.

Inclusion Criteria for healthy volunteers :

* Age ≥ 18 years ≤ 80 years
* Persons capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol. Written informed consent and any required authorisation must be obtained from the healthy volunteer prior to carrying out any procedure related to the protocol, including examinations to assess the eligibility of the person
* Persons who are affiliated to or are beneficiaries of a social security scheme according to local requirements.

Exclusion Criteria for patients :

- Independent physical activity exceeding INCa recommendations: Moderate physical activity greater than or equal to 300 minutes/week (≥5h) or intense physical activity greater than or equal to 150 minutes/week (≥2.5h)).

* Specific diet and/or any lipid-lowering treatment within 15 days prior to randomisation.
* Metformin treatment within 15 days prior to randomisation.
* Any medical conditions or co-morbidities likely to contraindicate the practice of physical activity. The list below is not exhaustive:

Previous stroke Myocardial infarction in the 6 months prior to inclusion Uncontrolled arterial hypertension Severe cardiovascular or respiratory disease Rheumatological/orthopaedic conditions or bone lesions at risk of fracture

* Presence of symptomatic cerebral metastasis(es).
* Prognosis estimated at less than 3 months.
* Unable to undergo medical monitoring of the trial and the various visits for geographical, social or psychological reasons.
* Persons deprived of their liberty or under guardianship (including curatorship).
* Pregnant or breast-feeding women (pregnancy test compulsory at inclusion).
* The patient does not have internet access / a smartphone / does not wish to download the AXOMOVE application required to take part in the study.

Exclusion Criteria for healthy volunteers :

* Patients with a history of cancer other than basal cell cancer, or who have already received systemic anti-cancer treatment.
* Persons with a special diet, metformin treatment and/or any lipid-lowering treatment in the 15 days prior to inclusion.
* Persons with moderate physical activity exceeding 300 minutes/week or intense physical activity exceeding 150 minutes/week.
* Persons deprived of their liberty or under guardianship (including curatorship).
* Pregnant or breast-feeding women (pregnancy test compulsory at inclusion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of adapted physical activity on the concentration of complex lipids in a population of patients with metastatic colorectal cancer treated with chemotherapy. | For 8 weeks
  The concentrations of complex lipids will be measured by high-performance liquid chromatography-mass spectrometry and by gas chromatography-mass spectrometry.
  The different concentrations of complex lipids will be compared between the 3 groups of patients (groups 1, 2 and 3) benefiting from a different frequency of adapted physical activity sessions.

SECONDARY OUTCOMES:
Evaluating and comparing adverse events linked to adapted physical activity | 24 months
  Safety will be assessed in the 3 physical activity groups according to NCI-CTCAE version 5.1
Evaluate and compare changes in patients' quality of life | During 8 weeks
  Quality of life will be assessed in the 3 physical activity groups by the quality of life questionnaire (FACT-C) at inclusion, at 4 weeks and at the end of 8 weeks of physical activity follow-up. This questionnaire is numbered from 0 to 4 (0 is the best case / 4 is the worst case).
  This questionnaire informe on the physical well-being, familial well-being, emotional well-being, functional well-being.
Prospective collection of biological plasma samples | During 8 weeks
  All samples are kept in order to analyze the expression of a marker of interest in a subpopulation of immune cells not included in the study panels a posteriori.
Progression-free survival | 24 months
  Disease response will be described at each evaluation.
Overall survival | 24 months
  Overall survival will be defined as the time elapsed between inclusion and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Julie VINCENT, Principal Investigator — Centre Georges François Leclerc
Locations (2):
- France (2):
  - Centre Georges-François Leclerc, Dijon
  - CHU Dijon (clinical investigation centre), Dijon

IPD SHARING:
Plan to Share IPD: No